CLINICAL TRIAL: NCT03951025
Title: Study of the Bioavailability of a Food Supplement Rich in Melatonin Administered Sublingually Compared to Its Oral Administration. Randomized, Crossover, Single-blind Study
Brief Title: Study of the Bioavailability of a Food Supplement Rich in Melatonin Administered Sublingually and Orally (MELATONIN)
Acronym: MELATONIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Fundació Eurecat (Other); Hospital Universitari Sant Joan de Reus (Other); Plantas Medicinales y Complementos Alimenticios (PLAMECA), S.A. (Unknown); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MELATONIN
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Biological Availability
Keywords: melatonin; oral administration; sublingual administration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin oral administration (Active Comparator): Consumption of one tablet with 1 mg of melatonin orally
  Interventions: Dietary Supplement: Melatonin oral administration
- Melatonin sublingual administration (Experimental): Consumption of one tablet with 1 mg of melatonin sublingually
  Interventions: Dietary Supplement: Melatonin sublingual administration

INTERVENTIONS:
Dietary Supplement: Melatonin oral administration — One tablet with1 mg of melatonin and 82 mg of excipients
  Arms: Melatonin oral administration
Dietary Supplement: Melatonin sublingual administration — One tablet with 1 mg of melatonin and 82 mg of excipients
  Arms: Melatonin sublingual administration

SUMMARY:
Sleep disorders represent an important public health problem that cause important personal problems, absenteeism and considerable health costs. Although the main drugs used for the treatment of insomnia are still Benzodiazepines and Z-drugs (Zolpidem, Zopiclone, Zaleplon), these are not entirely effective and have numerous side effects that lead to poor compliance with therapy . For the treatment of sleep disorders, alternative non-pharmacological therapies have also been implemented, such as cognitive therapy, relaxation therapy, and the introduction of new agents, including the use of melatonin as a human endogenous molecule with low or zero toxicity.

In Europe, the European Food Safety Authority (EFSA) has stated that "A cause and effect relationship is established between the consumption of melatonin and the alleviation of subjective feelings of jet lag. In order to present the declaration of health, the dose of melatonin should be between 0.5 and 5 mg and should be taken close to bedtime on the first day (and subsequent days) of the trip and the following days after arrival at destination.The target population is the general population ". On the other hand, the EFSA states that "A cause and effect relationship is established between the consumption of melatonin and the reduction of sleep onset latency. The Panel considers that to obtain the declared effect, 1 mg of melatonin should be consumed near bedtime. The target population is the general population."

The results of several studies in humans show that melatonin administered orally has a low bioavailability (approximately percentage) and a very short half-life. Therefore, it has been suggested that the sublingual route represents an attractive alternative for the administration of compounds that have a low bioavailability, since through this route, the substances are distributed throughout the body avoiding the loss of the compounds by their first-pass metabolism by the liver, as well as the loss by the process of absorption by the digestive system.

On this basis the present hypothesis is posed: the administration of melatonin sublingually will have a greater bioavailability than the administration of melatonin orally.

The main objective of this study was to quantify the bioavailability of 1 mg of melatonin when administered sublingually and orally.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age.
2. Firm the informed consent.

Exclusion Criteria:

1. Take supplements or multivitamin supplements or phytotherapeutic products that interfere with the treatment under study up to 30 days before the start of the study.
2. Present intolerances and / or food allergies related to melatonin.
3. Presenting anemia (hemoglobin ≤ 13 g/dL in men and ≤ 12 g/dL in women).
4. Being pregnant or intending to become pregnant.
5. Be in breastfeeding period.
6. Be a smoker
7. Participate in or have participate in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Bioavailability of melatonin calculated by the Area Under The Curve (AUC) | At week 1 and week 2. The extraction and bleeding points of melatonin will be at basal time, before taking the tablet and at 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours and 6 hours after tablet intake.
  Fasting melatonin blood levels will be determined before consuming the melatonin supplement until 6 hours postprandially at 7 points after consuming the melatonin supplement.
  The melatonin levels in plasma will be quantified with a Liquid Chromathography (LC)-(ESI+)- Mass Spectrometry (MS)/MS from their pure commercial standard using melatonin-d4 as internal standard.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | At week 1 and week 2. The extraction and bleeding points of melatonin will be at basal time, before taking the tablet and at 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours and 6 hours after tablet intake.
  Maximum plasma concentration of melatonin. Cmax will be measured by pharmacokinetics formulas from the melatonin values measured at different times (basal and postprandial)
Time for maximum plasma concentration (Tmax) | At week 1 and week 2. The extraction and bleeding points of melatonin will be at basal time, before taking the tablet and at 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours and 6 hours after tablet intake.
  Time period for the maximum plasma concentration of melatonin.
Half-life (T1/2) | At week 1 and week 2. The extraction and bleeding points of melatonin will be at basal time, before taking the tablet and at 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours and 6 hours after tablet intake.
  Time taken for half the initial dose of melatonin administered to be eliminated from the body
Melatonin urine levels | At week 1 and week 2. Urine at basal time and at 3 hours and 6 hours after tablet consumption.
  Determination of melatonin and/or its main metabolite 6-sulfatoxymelatonin in urine

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — Centro Tecnológico de Nutrición y Salud (Eurecat_Reus). Reus, Tarragona, Spain.
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No